CLINICAL TRIAL: NCT04621877
Title: Lay-Delivered Behavioral Activation in Senior Centers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); University of South Florida (Other); Weill Medical College of Cornell University (Other)
Responsible Party: Principal Investigator, Patrick Raue, Professor, School of Medicine: Psychiatry: Population Health, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00011434; R01MH124975 (NIH)
Record Dates: First submitted 2020-11-03; First posted 2020-11-09 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Volunteer-delivered Behavioral Activation - "Do More, Feel Better" (Experimental): "Do More, Feel Better" (DMFB) is a streamlined, simplified version of Behavioral Activation (BA) delivered by lay volunteers to depressed senior center clients.
  Interventions: Behavioral: Volunteer-delivered Behavioral Activation
- Master's Level Clinician-delivered Behavioral Activation (Active Comparator): Traditional Behavioral Activation (BA) delivered by master's level mental health clinicians
  Interventions: Behavioral: Master's level clinician-delivered Behavioral Activation

INTERVENTIONS:
Behavioral: Volunteer-delivered Behavioral Activation — Behavioral Activation as delivered by trained volunteers
  Arms: Volunteer-delivered Behavioral Activation - "Do More, Feel Better"
Behavioral: Master's level clinician-delivered Behavioral Activation — Behavioral Activation as delivered by trained master's level clinicians
  Arms: Master's Level Clinician-delivered Behavioral Activation

SUMMARY:
In response to large numbers of senior center clients who suffer untreated depression and the dearth of geriatric mental health providers, the investigators have simplified Behavioral Activation to be delivered by lay volunteers ("Do More, Feel Better"; DMFB). The focus of Behavioral Activation is to guide clients to reengage in daily pleasant and rewarding activities, and reduce depressive symptoms. If the investigators can show that the lay delivery model has positive impact in comparison to MSW-delivered Behavioral Activation, the investigators will have identified an effective intervention that can be used by a large untapped workforce of older adult volunteers across the nation.

DETAILED DESCRIPTION:
This Collaborative R01 application (UW, Cornell, USF) proposes to conduct an effectiveness trial of lay-delivered Behavioral Activation ("Do More, Feel Better"; DMFB), in comparison to MSW-delivered Behavioral Activation (MSW BA), for depressed (PHQ-9>10 and Ham-D>14) older (60+) senior center clients. The primary aim tests the effectiveness of DMFB, in comparison to MSW BA, on increasing overall activity level (target) and reducing depression symptoms. The investigators will test whether increased activity level predicts greater reduction in depression severity and whether increased activity's impact on depression is non-inferior across conditions. Secondarily, the investigators will test hypotheses associated with overall functioning, satisfaction with treatment, and client-level moderators. Lastly the investigators will explore longer-term client outcomes, delivery cost, and preparing for sustainability by exploring client, provider, and center factors related to intervention fidelity.

ELIGIBILITY:
Client Participants (anticipated enrollment: 288)

Inclusion Criteria:

Referral to study (stage 1):

1. Age ≥ 60 years.
2. Attends one of 18 participating Seattle, NYC, or Tampa area senior centers.
3. Patient Health Questionnaire (PHQ-9) score of ≥10 via routine screening.

Research assessment (stage 2):

1. Clinically-assessed HAM-D>14
2. Mini-Mental Status Exam (MMSE) ≥ 24 OR modified Telephone Interview for Cognitive Status (mTICS) ≥ 19
3. Off antidepressants or on a stable dose for 12 weeks.
4. Capacity to provide written consent for both research assessment and the BA intervention.

Client Participants Exclusion Criteria:

1. Current active suicidal ideation.
2. Presence of psychiatric diagnoses other than unipolar, non-psychotic major depression or generalized anxiety disorder by SCID-V (Structure Clinical Interview for DSM-V).
3. Severe or life-threatening medical illness (e.g., end stage organ failure).
4. Inability to speak English or Spanish

Volunteer Participants (anticipated enrollment: 36) Inclusion Criteria

1. Age ≥ 60 years.
2. Attends one of the participating Seattle, NYC, or Tampa-area senior centers.

Volunteer Participants Exclusion Criteria

1. Current major depressive disorder, alcohol or substance abuse, or manic, hypomanic, or psychotic symptoms (SCID-V);
2. Mini-Mental Status Exam (MMSE) ≥ 24 OR modified Telephone Interview for Cognitive Status (mTICS) ≥ 19;
3. Inability to speak and read English or Spanish

Clinician Participants (anticipated enrollment: 36) Inclusion Criteria

1. Master's degree in social work, counseling, marriage/family, or other clinical mental health degree
2. English or Spanish Speaking
3. Capacity to provide consent for all study procedures
4. Willing to audio record study sessions for supervision and evaluation

Clinician Participants Exclusion Criteria

1. Non-English or Non-Spanish speaking
2. Does not hold a Master's degree in social work, counseling, marriage/family, or other clinical mental health degree
3. Unable to provide consent
4. Unwilling to audio record study sessions for supervision and evaluation

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Estimated)
Dates: Start 2021-01-27 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Hamilton Rating Scale for Depression (HAM-D) | Change from Baseline HAM-D at 3, 6, 9, 24, and 36 weeks after treatment starts
  The HAM-D will be used as measure of depressive symptom severity. The HAM-D is a clinically administered measure and has been validated in a variety of psychiatric populations.
Behavioral Activation Scale (BADS) | Change from Baseline BADS at 3, 6, 9, 24, and 36 weeks after treatment starts
  The BADS will be used as the primary target measure, and yields a total score reflecting level of engagement in reinforcing activities. The BADS has shown good psychometric properties; studies have validated the BADS as a mechanism by which behavioral activation interventions reduces depression.

SECONDARY OUTCOMES:
World Health Organization Disability Assessment Schedule (WHODAS II) | Change from Baseline WHODAS-II at 3, 6, 9, 24, and 36 weeks after treatment starts
  The World Health Organization Disability Assessment Schedule II (WHODAS II)-12 item form will be used to assess overall functioning. This instrument is cross-culturally applicable and treats all disorders at parity when determining level of functioning. The WHODAS II assesses 6 domains: a. understanding and communicating; b.
  getting around; c. self-care; d. getting along with others; e. household and work activities; and f. participation in society. Each domain has factor loading of at least 0.70 and the items also load on a general disability factor which will be used in this proposal.
Client Satisfaction with Treatment (CSQ)- 3 Item | Administered at 3, 6, and 9 weeks after treatment starts
  The 3-item version of the Client Satisfaction Questionnaire (CSQ) will be used as a patient self-report measure of satisfaction with study interventions. The CSQ has high internal consistency and successfully distinguishes degrees of satisfaction even at the high end.

OTHER OUTCOMES:
Intervention Fidelity | Weekly for 9 weeks of treatment
  The "Do More, Feel Better" and BADT-R fidelity forms will be used by external raters to assess each interventionist's fidelity to the respective treatment modality. Global scores range from 0-6, with scores >3 indicating satisfactory levels of fidelity.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick J Raue, PhD, Principal Investigator — University of Washington
Locations (25):
- United States (25):
  - Brandon Senior Center, Brandon, Florida
  - Gardenville Dining & Activity Center, Gibsonton, Florida
  - Ruskin Senior Center, Ruskin, Florida
  - JL Young Apartments (Senior Housing), Tampa, Florida
  - Oaks at Riverview Senior Center, Tampa, Florida
  - Jewish Towers Senior Housing, Tampa, Florida
  - Town 'n Country Senior Center, Tampa, Florida
  - Progress Village Senior Center, Tampa, Florida
  - Diana Jones Senior Center, Brooklyn, New York
  - Edie Windsor SAGE Center, New York, New York
  - Hudson Guild Senior Center, New York, New York
  - Lincoln Square Senior Center, New York, New York
  - Goddard Riverside Community Center and NORC, New York, New York
  - Carver Senior Center, New York, New York
  - Dyckman Senior Center, New York, New York
  - Stanley M. Isaacs Neighborhood Center, New York, New York
  - SAGE Center Brooklyn at Stonewall House, New York, New York
  - Enumclaw Senior Center, Enumclaw, Washington
  - Greenwood Senior Center, Seattle, Washington
  - West Seattle Senior Center, Seattle, Washington
  - Southeast Seattle Senior Center, Seattle, Washington
  - GenPride Senior Center, Seattle, Washington
  - Casa Latina, Seattle, Washington
  - Centro de la Raza, Seattle, Washington
  - Pt Defiance Senior Center, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: Yes
We will deposit participant data into the NIMH informatics infrastructure (e.g., National Data Archive) to enable sharing of clinical research data.

REFERENCES:
- [Derived] Raue PJ, Sirey JA, Gum A, Hawrilenko M, Fisher DM. Protocol for a collaborative randomised effectiveness trial of lay-delivered versus clinician-delivered behavioural activation in senior centres. BMJ Open. 2022 Aug 23;12(8):e066497. doi: 10.1136/bmjopen-2022-066497. PMID 35998966